CLINICAL TRIAL: NCT00300703
Title: Ontario Prehospital Advanced Life Support (OPALS) Study Cardiac Arrest Database
Brief Title: OPALS Cardiac Arrest Database (OCAD)
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institute for Health Information (Other)
Responsible Party: Dr Ian Stiell, Ottawa Hospital Research Institute
Other Study IDs: 19975760-01H
Record Dates: First submitted 2005-09-13; First posted 2006-03-09 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To provide the infrastructure to answer prehospital research questions posed by scientists at academic health science centers and policy makers at multiple levels of government.

DETAILED DESCRIPTION:
To provide the infrastructure to answer prehospital research questions posed by scientists at academic health science centers and policy makers at multiple levels of government

ELIGIBILITY:
Inclusion Criteria:

* Ages 16 years and above

Exclusion Criteria:

under 16 yrs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * Ages 16 years and above
  Exclusion Criteria:
  under 16 yrs
Sampling Method: Probability Sample
Enrollment: 1538 (Actual)
Dates: Start 2006-01; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — OHRI
Locations (11):
- Canada (11):
  - Cambridge Base Hosptial, Cambridge, Ontario
  - Sudbury Base Hospital, Greater Sudbury, Ontario
  - Kingston Base Hosptial, Kingston, Ontario
  - London Base Hospital, London, Ontario
  - Halton Base Hosptial, Mississauga, Ontario
  - Niagara Falls Base Hospital, Niagara Falls, Ontario
  - Ottawa Base Hospital, Ottawa, Ontario
  - Peterborough Base Hospital, Peterborough, Ontario
  - Lambton Base Hospital, Sarnia, Ontario
  - Thunder Bay Base Hospital, Thunder Bay, Ontario
  - Windsor Base Hospital, Windsor, Ontario